CLINICAL TRIAL: NCT02977780
Title: INdividualized Screening Trial of Innovative Glioblastoma Therapy (INSIGhT)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Patrick Wen, MD (Other)
Collaborators: Eli Lilly and Company (Industry); Celgene (Industry); Puma Biotechnology, Inc. (Industry); Accelerate Brain Cancer Cure (Other); Quadriga Biosciences, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Patrick Wen, MD, Director, Center for Neuro-Oncology, Dana-Farber Cancer Institute
Organization: Dana-Farber Cancer Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16-443
Record Dates: First submitted 2016-11-18; First posted 2016-11-30 (Estimated); Last update posted 2025-11-10 (Actual); Status verified 2025-10

CONDITIONS: Glioblastoma
Keywords: Glioblastoma
MeSH Terms: conditions — Glioblastoma | interventions — Temozolomide; neratinib; abemaciclib; 1-ethyl-7-(2-methyl-6-(1H-1,2,4-triazol-3-yl)pyridin-3-yl)-3,4-dihydropyrazino(2,3-b)pyrazin-2(1H)-one

STUDY DESIGN:
Intervention Model Description: This research study is studying several investigational drugs as a possible treatment for Glioblastoma (GBM).
  The drugs involved in this study are:
  Abemaciclib: start date= 12/9/2017 Temozolomide (temodar): start date= 12/9/2017 Neratinib: start date= 12/9/2017 CC115: start date= 12/9/2017 QBS10072S: start date= 12/13/2022
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Temozolomide (Active Comparator): * Daily Radiation for a maximum of 49 days.
  * Temozolomide will be administered orally on a daily dosing schedule
  * Temozolomide will be administered approximately 2-3 hours before each session of radiotherapy
  * Temozolomide will also be administered post radiation for up to 6 cycles (5 days/cycle)
  Interventions: Drug: Temozolomide
- Neratinib with Temozolomide (Experimental): * Daily Radiation for a maximum of 49 days.
  * Temozolomide will be administered orally on a daily dosing schedule
  * Temozolomide will be administered approximately 2-3 hours before each session of radiotherapy
  * Neratinib will be taken post radiation at a daily oral pre-determine dose
  Interventions: Drug: Temozolomide; Drug: Neratinib
- QBS10072S (Experimental): Daily Radiation for a maximum of 49 days.
  QBS10072S will be administered on Day 1 of Radiation Treatment
  QBS10072S will be administered post- radiation for up to 6 cycles
  Interventions: Drug: QBS10072S
- Abemaciclib with Temozolomide (Experimental): * Daily Radiation for a maximum of 49 days.
  * Temozolomide will be administered orally on a daily dosing schedule during radiation
  * Temozolomide will be administered approximately 2-3 hours before each session of radiotherapy
  * Abemaciclib will be taken post radiation at a twice daily oral pre-determined dose
  Interventions: Drug: Temozolomide; Drug: Abemaciclib
- CC-115 (Experimental): * Twice daily oral dosing of CC-115
  * Daily Radiation for a maximum of 49 days
  * CC115 will also be taken twice daily post radiation
  Interventions: Drug: CC-115

INTERVENTIONS:
Drug: Temozolomide — Temzolomide capsules
  Other Names: Temodar
  Arms: Abemaciclib with Temozolomide; Neratinib with Temozolomide; Temozolomide
Drug: Neratinib — Neratinib tablets
  Arms: Neratinib with Temozolomide
Drug: QBS10072S — QBS10072S administered intravenously
  Arms: QBS10072S
Drug: Abemaciclib — Abemaciclib tablets
  Arms: Abemaciclib with Temozolomide
Drug: CC-115 — CC-115 tablets
  Arms: CC-115

SUMMARY:
This research study is studying several investigational drugs as a possible treatment for Glioblastoma (GBM).

The drugs involved in this study are :

* Abemaciclib (arm is currently closed to accrual)
* Temozolomide (temodar)
* Neratinib (arm is currently closed to accrual)
* CC115 (arm is currently closed to accrual)
* QBS10072S

DETAILED DESCRIPTION:
This research study is a Phase II clinical trial. Phase II clinical trials test the safety and effectiveness of an investigational drug to learn whether the study drug works in treating a specific disease. "Investigational" means that the drug is being studied.

In this research study, the investigators are looking to compare the effects, good and bad, of the standard of care with the three investigational agent sub-studies Abemaciclib, Neratinib, CC115, QBS10072S to help people with Glioblastoma including the specific molecular changes in the genes and proteins.

The FDA has approved Temozolomide (temodar) as a treatment for this disease, however the FDA has not approved Abemaciclib, CC115, Neratinib, QBS10072S for any diseases.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have histologically confirmed intracranial glioblastoma or gliosarcoma following maximum surgical resection. Tumors primarily localized in the infratentorial compartment will be excluded.
* Participants may have had prior surgery for glioblastoma or gliosarcoma but no systemic or radiation therapy.
* Age ≥ 18 years.
* Karnofsky performance status ≥60
* Participants must have normal organ and marrow function as defined below:

  * Leukocytes ≥3,000/mL
  * Absolute neutrophil count ≥1,500/mL
  * Platelets ≥100,000/mL
  * Hemoglobin ≥ 9g/dl
  * Total bilirubin within normal institutional limits (except for participant's with Gilbert's disease)
  * AST(SGOT)/ALT(SGPT) ≤ 2.5 × institutional upper limit of normal
  * Creatinine ≤ institutional upper limit of normal OR
  * Creatinine clearance ≥ 60 mL/min/1.73 m2 for participants with creatinine levels above institutional normal.
  * Potassium within normal institutional range, or correctable with supplements
  * Serum amylase ≤ 1.5 x institutional upper limit of normal
  * Serum lipase ≤ 1.5 x institutional upper limit of normal
  * INR < 2.0
  * PTT ≤ institutional upper limit of normal, unless receiving therapeutic low molecular weight heparin
* Must be able to swallow pills.
* Participants must plan to begin radiation therapy 14-42 days after surgical resection.
* Immunohistochemically negative for IDH1 R132H mutation.
* Evidence that the tumor MGMT promoter is unmethylated by standard of care assays.
* Genotyping data available or in process (data must be available at time of initial registration if randomization probabilities differ across biomarker subgroups as determined by the DFCI Coordinating Center) to assign biomarker subgroups through whole exome sequencing, whole genome copy number analysis, or a combination as described in Section 9.1.
* MRI with gadolinium should be obtained within 21 days prior to beginning treatment. Patients without measurable disease are eligible. Participants must be able to undergo MRIs (CTs are not allowed for response assessment on study).
* The effects of the experimental agents used in this study on the developing human fetus are unknown. For this reason and because other therapeutic agents used in this trial are known to be teratogenic, women of child-bearing potential (women who are not free from menses for > 2 years, post hysterectomy/oophorectomy, or surgically sterilized) and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation unless otherwise specified in sub-study that the participant is randomized to. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.
* For women of child bearing potential (women who are not free from menses for > 2 years, post hysterectomy/oophorectomy, or surgically sterilized) a negative serum pregnancy test must be documented prior to initial registration.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Participants will not be eligible if the original diagnosis was a lower grade glioma and a subsequent histologic diagnosis revealed glioblastoma.
* Planned major surgery.
* Participants who are receiving any other investigational agents.
* Participants who have had any prior cranial radiotherapy.
* Planned use of Optune™.
* History of a different malignancy, unless (a) have been disease-free for at least 2 years and are deemed by the investigator to be at low risk for recurrence of that malignancy, and/or (b) malignancy was cervical cancer in situ, superficial bladder cancer or basal cell or squamous cell carcinoma of the skin, and malignancy has been treated. Patients who meet the above listed criteria and are only on preventative treatment will be deemed eligible.
* History of intratumoral or peritumoral hemorrhage if deemed significant by the treating physician.
* Impaired cardiac function or clinically significant cardiac diseases, including any of the following:
* Active uncontrolled cardiac disease, including cardiomyopathy, congestive heart failure (New York Heart Association functional classification of ≥2), unstable angina, myocardial infarction within 12 months of enrollment, or ventricular arrhythmia.
* Known history of congenital QT prolongation or Torsade de pointes (TdP).
* Complete left bundle branch or bifascicular block.

  --QTc interval > 450 ms for men or > 470 ms for women.
* Persistent or history of clinically meaningful ventricular arrhythmias or atrial fibrillation.
* Unstable pectoris or myocardial infarction ≤ 3 months prior to starting study treatment.
* Uncontrolled hypertension (blood pressure ≥ 160/95 mmHg).
* Other clinically significant heart disease such as congestive heart failure requiring treatment.
* Uncontrolled diabetes mellitus, or subjects with either of the following:
* Fasting blood glucose (FBG defined as fasting for at least 8 hours) ≥ 200 mg/dL (7.0 mmol/L), or
* HbA1c ≥ 8%
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, chronic liver disease (e.g., cirrhosis, hepatitis), chronic renal disease, pancreatitis, chronic pulmonary disease, or psychiatric illness/social situations that would limit compliance with study requirements. Subjects must be free of any clinically relevant disease (other than glioma) that would, in the treating investigator's opinion, interfere with the conduct of the study or study evaluations.
* Known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNS [qualitative] is detected).
* Known acute or chronic pancreatitis.
* Participants with active diarrhea ≥ CTCAE grade 2 despite medical management.
* Active infection requiring antibiotics.
* Pregnant or breastfeeding.
* Impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of study drug (e.g., ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, or extensive small bowel resection). Participants with unresolved diarrhea ≥ CTCAE grade 2 will be excluded as previously indicated.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to any of the experimental agents or other agents used in study.
* Participants taking an enzyme-inducing anti-epileptic drug (EIAED): phenobarbital, phenytoin, fosphenytoin, primidone, carbamazepine, oxcarbazepine, eslicarbazepine, rufinamide, and felbamate. Participant must be off any EIAEDs for at least 7 days prior to planned start of study treatment. A list of EIAED and other inducers of CYP3A4 is provided. Among non-EIAED, caution is recommended with use of valproic acid due to potential for drug interaction.
* Participants taking a drug known to be strong inhibitors or inducers of isoenzyme CYP3A. Participant must be off CYP3A inhibitors and inducers for at least 7 days prior to planned start of study treatment. NOTE: participants must avoid consumption of Seville orange (and juice), grapefruit or grapefruit juice, grapefruit hybrids, pummelos and exotic citrus fruits from 7 days prior to planned start of study treatment and during the entire study treatment period due to potential CYP3A4 interaction.
* Current use of herbal preparations/medications, including but not limited to: St. John's wort, Kava, ephedra (ma huang), gingko biloba, dehydroepiandrosterone (DHEA), yohimbe, saw palmetto, ginseng. Participants should stop using these herbal medications 7 days prior to planned start of study treatment.
* Current use of warfarin sodium or any other coumadin-derivative anticoagulant. Participant must be off Coumadin-derivative anticoagulants for at least 7 days prior to planned start of study treatment. Low molecular weight heparin and factor Xa inhibitors are allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 460 (Estimated)
Dates: Start 2017-02-09 (Actual); Primary Completion 2028-02-01 (Estimated); Study Completion 2028-04-30 (Estimated)

PRIMARY OUTCOMES:
Overall Survival in Experimental Arms Compared with Standard Therapy | 2 years

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | 2 years
  Safety will be assessed by quantifying the toxicities and grades experienced by subjects, including serious adverse events (SAEs). The following will also be measured as part of safety: laboratory safety assessments, KPS status, vital signs and physical examinations.
Progression Free Survival Among Experimental Arms And Biomarker Groups | 2 years
Overall Survival Among Experimental Arms And Biomarker Groups | 2 years
Association Between Progression Free Survival and Overall Survival Effects Of Experimental Agents | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Y Wen, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (12):
- United States (12):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Columbia University Medical Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Cleveland Clinic, Cleveland, Ohio
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Lifespan / Rhode Island Hospital, Providence, Rhode Island
  - UT MD Anderson Cancer Center, Houston, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - University of Virginia Health System, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rahman R, Trippa L, Lee EQ, Arrillaga-Romany I, Fell G, Touat M, McCluskey C, Wiley J, Gaffey S, Drappatz J, Welch MR, Galanis E, Ahluwalia MS, Colman H, Nabors LB, Hepel J, Elinzano H, Schiff D, Chukwueke UN, Beroukhim R, Nayak L, McFaline-Figueroa JR, Batchelor TT, Rinne ML, Kaley TJ, Lu-Emerson C, Mellinghoff IK, Bi WL, Arnaout O, Peruzzi PP, Haas-Kogan D, Tanguturi S, Cagney D, Aizer A, Doherty L, Lavallee M, Fisher-Longden B, Dowling S, Geduldig J, Watkinson F, Pisano W, Malinowski S, Ramkissoon S, Santagata S, Meredith DM, Chiocca EA, Reardon DA, Alexander BM, Ligon KL, Wen PY. Inaugural Results of the Individualized Screening Trial of Innovative Glioblastoma Therapy: A Phase II Platform Trial for Newly Diagnosed Glioblastoma Using Bayesian Adaptive Randomization. J Clin Oncol. 2023 Dec 20;41(36):5524-5535. doi: 10.1200/JCO.23.00493. Epub 2023 Sep 18. PMID 37722087
- [Derived] Groot J, Ott M, Wei J, Kassab C, Fang D, Najem H, O'Brien B, Weathers SP, Matsouka CK, Majd NK, Harrison RA, Fuller GN, Huse JT, Long JP, Sawaya R, Rao G, MacDonald TJ, Priebe W, DeCuypere M, Heimberger AB. A first-in-human Phase I trial of the oral p-STAT3 inhibitor WP1066 in patients with recurrent malignant glioma. CNS Oncol. 2022 Jun 1;11(2):CNS87. doi: 10.2217/cns-2022-0005. Epub 2022 May 16. PMID 35575067

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-12-04): https://cdn.clinicaltrials.gov/large-docs/80/NCT02977780/Prot_SAP_000.pdf